CLINICAL TRIAL: NCT03349944
Title: Effect of High Intensity Interval Training on Nuclear Orphan Receptor Expression and Adrenergic Signaling in Skeletal Muscle of Persons With Type 2 Diabetes.
Brief Title: Effect of Training Intensity on Health Outcomes in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Morten Hostrup, PhD (Other)
Responsible Party: Sponsor-Investigator, Morten Hostrup, PhD, Assistant Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NOR
Record Dates: First submitted 2017-11-17; First posted 2017-11-22 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate intensity training (Active Comparator): Moderate continuous exercise three times pr. week for 50 min.
  Interventions: Behavioral: Training
- High intensity training (Experimental): High intensity interval training three times pr. week for 15 min.
  Interventions: Behavioral: Training

INTERVENTIONS:
Behavioral: Training — The duration of the training intervention is 10 weeks of either moderate exercise og high intensity interval training.

SUMMARY:
The project will investigate high intensity interval training on the glucose regulation in type 2 diabetic subjects compared to moderate continuous exercise.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetes Age: 30-70 Non smokers (minimum the last 15 years) Inactive lifestyle (<2 hours pr. week) BMI <35 kg/m2

Exclusion Criteria:

Smoking Prior cardiavascular diseases Alcohol intake 14> units pr. week.

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
HbA1c | From baseline measure to post test: 10 weeks
  Long term blood glucose levels

SECONDARY OUTCOMES:
Oral glucose tolerance test | From baseline measure to post test: 10 weeks
  75gr glucose is ingested, bllod sampling over the following two hours

CONTACTS AND LOCATIONS:
Locations (1):
- August Krogh Building, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Baasch-Skytte T, Gunnarsson TP, Fiorenza M, Bangsbo J. Skeletal muscle proteins important for work capacity are altered with type 2 diabetes - Effect of 10-20-30 training. Physiol Rep. 2021 Jan;9(1):e14681. doi: 10.14814/phy2.14681. PMID 33426802